CLINICAL TRIAL: NCT04752501
Title: Maladaptive Psychosocial Beliefs and Adolescents With Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Mitchell Selhorst, Principal Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB18-00724.2
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Patellofemoral Pain Syndrome; Knee Pain Chronic; Patellofemoral Syndrome; Anterior Knee Pain Syndrome
Keywords: Knee; Adolescent; Psychologically-informed; Anterior Knee Pain
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This research study is a blinded randomized controlled trial. The participants will not be made aware which education video series they watch is the control and which is the intervention. The study staff will be blinded to group allocation until after measurements are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychologically Informed Video Series (Experimental): This 3 part educational video series will teach participants how the body processes nociception and experiences pain, and pain does not mean tissues are being damaged. Additionally we will use the framework called the "Common Sense Model of Self-Regulation" which advocates for education to address five cognitive dimensions: (1) identity (the effort to evaluate symptoms and label the illness); (2) cause (the subjectively formulated belief of what is causing the symptoms); (3) time-line (the patient's perception of how long the problem will last); (4) consequences (the patient's predictions of how the illness will affect them in different areas of their life); and (5) controllability (the patient's belief regarding their outcome and personal ability to change it); Simple methods of cognitive restructuring; and how to respond to activity-related pain.
  Interventions: Other: Psychologically Informed Education
- Biomedical Education Video Series (Active Comparator): Participants in the control (biomedical education) group will watch a series videos on the iPad equal in length to the psychologically informed video series. The control video will discuss basic anatomy of the knee and provide no psychosocial education or positive reinforcement about their condition, basic strengthening exercises and proper lower extremity mechanics
  Interventions: Other: Biomedical Education (Control)

INTERVENTIONS:
Other: Psychologically Informed Education — This arm will provide an education intervention which will attempt to address maladaptive psychological behaviors in adolescents with knee pain
  Arms: Psychologically Informed Video Series
Other: Biomedical Education (Control) — This arm will provide education of basic knee anatomy, lower extremity mechanics, and simple exercises and will not address maladaptive psychological behaviors
  Arms: Biomedical Education Video Series

SUMMARY:
This is a randomized prospective study assessing the impact of psychosocial factors on pain and physical performance among adolescents with patellofemoral pain. A set of psychosocial surveys assessing fear avoidance beliefs, kinesiophobia, and pain catastrophizing will be completed by the participant/parents. Participants will then complete an activity questionnaire, numeric pain rating scale, and a self-report questionnaire of functional ability. Participants will then be randomized into one of two groups (psychologically informed education group and a control group). Participants will view a series of educational videos (based upon group assignment) and complete physical therapy exercises for lower extremity strengthening, flexibility, and neuromuscular control. Participants with patellofemoral pain will then complete follow-up surveys of their psychosocial beliefs, pain and self-reported functional ability through REDcap at immediately post-intervention, 1 week, 3 weeks, 6 weeks, and 3 months.

ELIGIBILITY:
Inclusion Criteria:

• Having patellofemoral pain as defined as: Pain around or behind the patella, which is aggravated by at least one activity that loads the patellofemoral joint during weight bearing on a flexed knee (e.g., squatting, stair ambulation, jogging/running, hopping/jumping).

Exclusion Criteria:

* Prior history of patellar dislocation.
* Suspicion of other diagnosis of the knee by evaluating physical therapist or principal investigator.
* Other concomitant injury of the leg.
* Prior history of knee surgery.
* Red flags present for non-musculoskeletal involvement (bowel/bladder problems, saddle anesthesia, progressive neurological deficits, recent fever or infection, unexplained weight loss, unable to change symptoms with mechanical testing).
* Numbness and tingling in any lumbar dermatome.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Change in Anterior Knee Pain Scale | Baseline, 1 week, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), and 3 months]
  Assessment of change of the Anterior Knee Pain Scale (AKPS). The AKPS is a self-reported 13 item questionnaire with discrete categories related to various levels of current knee function. Categories within each item are weighted, and responses are summed to provide an overall score of 0-100, with 100 representing no disability. The Anterior Knee Pain Scale is found to be valid and reliable in patients from 12-50 years of age presenting with anterior knee pain with a test-retest reliability of .95 (Watson, 2005). A change of 8-10 points represent the minimal clinical difference (Crossley, 2004).

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale | Baseline, 1 week, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), and 3 months]
  The Numeric Pain rating scale asks the patient their highest pain in the last 24 hours. The Numeric Pain Rating Scale is a 0-10 scale subjectively assessing a patients perceived level of pain. With 0 on the scale = to no pain, and 10 = to the worst pain imaginable. The use of the Numerical Pain Rating Scale for assessing pain has been validated for use in patients with knee pain and has been found to have a minimal detectable change of 1 points.
Change in self-reported physical activity level. | Baseline, 1 week, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), and 3 months]
  Change in Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Activity. PROMIS physical activity scale assesses activity over the past week. Each question has five response options ranging in value from 1 to 5. The responses are summed with scores ranging from 8-40 with 8 representing the lowest physical activity and 40 representing the highest physical activity. Raw scores are rescaled into a standardized T-score with a mean of 50 and a standard deviation (SD) of 10.
Change in Fear-Avoidance Beliefs | Baseline, 1 week, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), and 3 months]
  Change in fear avoidance beliefs as measure by the Fear Avoidance Beliefs Questionnaire Physical Activity scale (FABQ-PA). The FABQ-PA quantifies the patient's fear of pain and beliefs about avoiding activity. The FABQ-PA is a 5-item self-report measure which assesses an individual's fear-avoidance of painful activity and is modified for the knee. The FABQ-PA is modified by changing the word "back" to "knee" on the questionnaire. Each item is scored on a 0-6 scale, with 0 indicating completely disagree and 6 indicating completely agree. Questions 2-5 are summed to create a final score of 0-24, with high scores indicating higher fear avoidance beliefs.
Change in Kinesiophobia | Baseline, 1 week, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), and 3 months]
  Change in kinesiophobia beliefs as measure by the Tampa Scale for Kinesiophobia-11 scale. The TSK-11 is an 11-item questionnaire that assesses fear of injury due to movement. Patients are asked to make ratings of their degree of agreement with each of the 11 statements, for instance, 'Pain lets me know when to stop exercising so that I don't injure myself'. Ratings range from 1 (strongly disagree) to 4 (strongly agree). The responses are summed to yield a total score of 11-44 where higher values reflect higher kinesiophobia.
Change in Pain Catastrophizing | Baseline, 1 week, 3 weeks (18-24 days post-evaluation), 6 weeks (39-46 days post-evaluation), and 3 months]
  Change in pain catastrophizing as measured by the pain catastrophizing scale-child version (PCS-c). The PCS-c is a 13-item self-report measure designed to assess a child's pain catastrophizing. Each item is rated on a 5-point scale, ranging from 0 (not at all) to 4 (all the time). The responses are summed to yield a total score of 0-52 where higher values reflect higher pain catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Selhorst, DPT, PHD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital Sports and Ortho PT East Broad, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: As a part of this research, it will be necessary to collect identifying information. Even though the final dataset will be stripped of identifiers prior to release for sharing, the patient sample is composed of minors who are a protected patient population Thus, we will make the data and associated documentation available to users only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed. Aggregate data including sample means, standard deviations, frequencies and significance values will be shared through peer-reviewed publications and conference abstracts. Email requests for data-sharing agreements to Mitchell.Selhorst@Nationwidechildrens.org

REFERENCES:
- [Background] Grotle M, Garratt AM, Krogstad Jenssen H, Stuge B. Reliability and construct validity of self-report questionnaires for patients with pelvic girdle pain. Phys Ther. 2012 Jan;92(1):111-23. doi: 10.2522/ptj.20110076. Epub 2011 Oct 20. PMID 22016375
- [Background] Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. J Behav Med. 2016 Dec;39(6):935-946. doi: 10.1007/s10865-016-9782-2. Epub 2016 Aug 11. PMID 27515801
- [Background] Robins H, Perron V, Heathcote LC, Simons LE. Pain Neuroscience Education: State of the Art and Application in Pediatrics. Children (Basel). 2016 Dec 21;3(4):43. doi: 10.3390/children3040043. PMID 28009822
- [Background] Vlaeyen JWS, Linton SJ. Fear-avoidance model of chronic musculoskeletal pain: 12 years on. Pain. 2012 Jun;153(6):1144-1147. doi: 10.1016/j.pain.2011.12.009. Epub 2012 Feb 8. No abstract available. PMID 22321917
- [Background] Wang YC, Hart DL, Stratford PW, Mioduski JE. Baseline dependency of minimal clinically important improvement. Phys Ther. 2011 May;91(5):675-88. doi: 10.2522/ptj.20100229. Epub 2011 Mar 3. PMID 21372203
- [Background] Watson CJ, Propps M, Ratner J, Zeigler DL, Horton P, Smith SS. Reliability and responsiveness of the lower extremity functional scale and the anterior knee pain scale in patients with anterior knee pain. J Orthop Sports Phys Ther. 2005 Mar;35(3):136-46. doi: 10.2519/jospt.2005.35.3.136. PMID 15839307
- [Background] Crossley KM, Bennell KL, Cowan SM, Green S. Analysis of outcome measures for persons with patellofemoral pain: which are reliable and valid? Arch Phys Med Rehabil. 2004 May;85(5):815-22. doi: 10.1016/s0003-9993(03)00613-0. PMID 15129407
- [Derived] Selhorst M, Hoehn J, Schmitt L, Benedict J, Fernandez-Fernandez A. The Effect of a Psychologically Informed Video Series to Treat Adolescents With Patellofemoral Pain: A Randomized Controlled Trial. J Orthop Sports Phys Ther. 2023 Oct;53(10):634-642. doi: 10.2519/jospt.2023.12041. PMID 37706686